CLINICAL TRIAL: NCT04635722
Title: EMPOWER: Individualized Dietary Improvement Program
Brief Title: EMPOWER Weight Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Mindy Lee, Graduate Research Assistant, University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18069_Empower
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Obesity; Overweight; Weight Loss; Diet Habit
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Before and after study design with one interventional group and no control or placebo group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight Management Intervention (Experimental): During a 12-month period, participants will attend a total of 22 diet improvement sessions, each of which will last approximately 1 hour. Twelve sessions will be held in the first 5 months and will be focused on safe and efficient weight loss. The participants will learn to create a personalized weight loss diet from their kitchen based on their diet practice and food preference. The next 10 sessions will be held in the last 7 months and will be focused on weight maintenance and healthy eating. The participants will build skills to select foods and create meals that prevent them from overeating. Participants will be followed by daily self-weighing for 1 year after intervention.
  Interventions: Behavioral: Weight Management Intervention

INTERVENTIONS:
Behavioral: Weight Management Intervention — Participants attend group and individual dietary education sessions. Participants create a diet plan that satisfies their needs. Participants aim to lose 1 pound weekly until a BMI of 25 is reached. Participants are evaluated through daily self-weighing, dietary records, and food frequency questionnaires.

SUMMARY:
This research is to develop a virtual weight loss and weight maintenance program through dietary modifications for adults with obesity. Although scientific studies have shown the feasibility of rapid and safe dietary weight loss and subsequent weight maintenance, no efficacious dietary weight management program is widely available, and thus bariatric surgery remains the most reliable approach for weight loss/management. Safe and effective dietary weight loss and subsequent weight maintenance require flexible, individualized advice by an experienced dietitian/nutritionist.

DETAILED DESCRIPTION:
EMPOWER is a remote weight management program utilizing an online textbook platform, E-Text, and mobile web application. EMPOWER is a two-year program: 1-year intervention, 1-year follow up. Data is collected via FFQ (NIH DHQIII), daily weighing using a wifi-enabled scale, and 24-hour dietary records via the web application. EMPOWER consists of 19 online sessions (45 minutes/each) and 3 individual advising sessions with an RD.

EMPOWER aims to improve health parameters related to obesity, such as hyperlipidemia and hypertension. Health parameters will be monitored primarily by the subject's personal physician. Any test results will be sent to the EMPOWER research team for analysis via REDCap.

EMPOWER team consists of social workers in addition to nutrition experts. The social work team aims to monitor and improve lifestyle, stress management, and behavior.

ELIGIBILITY:
Inclusion Criteria:

* body mass index in the overweight or obese range (BMI) >28 kg/m2 (if Asian, BMI >25kg/m2);
* not currently pregnant or lactating;
* have Wi-Fi at home, a working email, and an iPhone or Android smartphone;
* self-reported obesity co-morbidities (such as diabetes type 2 or hyperlipidemia);
* be a Carle Foundation Hospital patient and have regular contact with a primary care physician;
* not using insulin injection;
* able to attend the 22 (1 hour) diet improvement sessions;
* willing and safe to lose 20 lb. or more for 6 months and maintain a healthy weight for one year;
* keep weighing their weight for two years;
* fluent in reading and writing English.

Exclusion Criteria:

* age <18 or >75 years;
* body mass index of <28 kg/m2 (if Asian, BMI <25kg/m2);
* currently pregnant;
* currently lactating;
* use insulin injection;
* not able to attend the 22 (1 hour) diet improvement sessions for 1 year;
* failed to set up a Wi-Fi scale;
* failed to submit a FFQ.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-08-11 (Estimated); Study Completion 2023-08-11 (Estimated)

PRIMARY OUTCOMES:
Body weight | Change from baseline (0 month) to 6 month, 12 month, 18 month, and 24 month
  Body weight in kilograms measured on a standard scale (Withings, US)

SECONDARY OUTCOMES:
Waist circumference | Change from baseline (0 month) to 6 month,12 month, 24 month
  Waist circumference in centimeters measured using a standard measuring tape
Hip circumference | Change from baseline (0 month) to 6 month, 12 month, 24 month
  Hip circumference in centimeters measured using a standard measuring tape
Body composition | Change from baseline (0 month) to 6 month, 12 month, 24 month
  Body fat measured using InBody 270
Body composition | Change from baseline (0 month) to 6 month, 12 month, 24 month
  lean mass measured using InBody 270
Protein Intake | Change from baseline (0 month) to 12 month
  Protein intake in grams and grams/100 kilo-calories using a food frequency questionnaire (FFQ)
Protein Intake | Periodically from baseline (0 month) to 12 month
  Protein intake in grams and grams/100 kilo-calories using a 24-hour record
Fiber Intake | Change from baseline (0 month) to 12 month
  Fiber intake in grams and grams/100 kilo-calories using a food frequency questionnaire (FFQ)
Fiber Intake | Periodically from baseline (0 month) to 12 month
  Fiber intake in grams and grams/100 kilo-calories using a 24-hour record
Health parameters as identified by subject's personal physician | As ordered by personal physician from baseline (0 month) to 24 months
  Tests may include but are not limited to CBC, CMP, Lipid panel
Blood pressure | Change from baseline (0 month) to 6 month, 12 month, 24 month
  Blood pressure measured as systolic/diastolic. Two measurements will be taken with subjects at rest. Measurements will be averaged.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No